CLINICAL TRIAL: NCT06278597
Title: Automatic Evaluation of the Anterior Chamber Angle Width by a New Non-contact Optical Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GLC02-22
Record Dates: First submitted 2024-02-15; First posted 2024-02-26 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: NACA Estimator — Grading of peripheral anterior chamber width with the Narrow Anterior Chamber Angle (NACA) Estimator

SUMMARY:
The aim of the study is to evaluate an objective, non-invasive optical device able to quantify, without eye contact, the width of the irido-corneal angle and to better identify cases of narrow angle or angle closure that may be prevented with relatively simple treatments.

DETAILED DESCRIPTION:
Worldwide, glaucoma has been identified as a leading cause of blindness, second only to cataract. The two most common types of glaucoma are primary open-angle and angle closure glaucoma (PACG), both characterized by progressive and irreversible degeneration of the retinal ganglion cells and axons. In PACG, the optic neuropathy occurs as a consequence of raised intraocular pressure (IOP) resulting from physical obstruction of aqueous outflow or degenerative changes in the trabecular meshwork. Angle closure is the result of an anatomic characteristic that causes closure of the drainage angle by synechial or appositional approximation between the iris and the trabecular meshwork, blocking access to aqueous humor. Although the most common mechanism responsible for angle closure is relative pupillary block, this is not the only one. Angle crowding can be caused by plateaus iris, or by multiple mechanisms such as choroidal thickness and uveal expansion.

A careful analysis of the anterior chamber angle is considered the main management strategy for PACG. The Van Herick grading of limbal anterior chamber depth is considered a screening tool for the estimation of angle width although gonioscopy remains the clinical reference standard for assessing the presence of narrow or closed angle. Ultrasound biomicroscopy, Scheimpflug imaging and anterior segment optical coherence tomography are considered as non-invasive alternatives to gonioscopy. However, these techniques are expensive and also have drawbacks. Therefore, there is a need for an easy and objective method able to evaluate the angle width for screening purposes in clinical practice.

Based on these findings, the purpose of the present study is to evaluate an objective, non-invasive optical device able to quantify, without eye contact, the width of the irido-corneal angle and to better identify cases of narrow angle or angle closure that may be prevented with relatively simple treatments.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate and ability to understand and sign an informed consent.
* 18 years of age or older.
* Healthy subjects, patients with PACS or angle closure as defined by the EGS Guidelines.
* The right eye will be included in the study for all patients, unless a clinical contraindication to the examination is present.

Exclusion Criteria:

* Inability to understand and sign an informed consent.
* Any prior ocular surgery or laser treatment with the potential to alter the natural anatomy of the anterior segment of the eye.
* Corneal or conjunctival abnormalities that preclude an adequate view of the anterior chamber.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Agreement between the automatic Narrow Anterior Chamber Angle Estimator grading of peripheral anterior chamber width with clinical grading as performed by Van Herick (VH) test at slit lamp | 12 months
  The angle is graded by the NACA estimator as the ratio between the peripheral anterior chamber depth and limbal-corneal thickness, as observed in the slit lamp by the microscope section. A high-resolution camera will synchronously acquire the images to generate the irido-corneal angle grade that will be classified in four grades following the VH classification.
  The standard VH grading scale will be:
  * 1 = space between iris and corneal endothelium of <¼ corneal thickness (angle closure likely),
  * 2 = space between iris and corneal endothelium of ¼ corneal thickness (angle closure possible),
  * 3 = space between iris and corneal endothelium of ½ corneal thickness (angle closure unlikely),
  * 4 = space between iris and corneal endothelium ≥ 1 (corneal thickness angle closure very unlikely).
Agreement between the automatic Narrow Anterior Chamber Angle Estimator grading of peripheral anterior chamber width with clinical grading as performed by gonioscopy. | 12 months
  The angle will be graded for each quadrant at gonioscopy using the modified Shaffer grading system, by which each grade corresponds to the visibility of the different angle structures.

SECONDARY OUTCOMES:
Reproducibility (intra-session) and repeatability (inter-session) of the peripheral anterior chamber width (PACW) evaluation by the Narrow Anterior Chamber Angle Estimator | 12 months
Sensitivity and specificity of NACA Estimator grading of PACW in detecting primary angle closure suspects as classified by clinical gonioscopy. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione GB Bietti, Roma, Italy, Italy

IPD SHARING:
Plan to Share IPD: No